CLINICAL TRIAL: NCT00219492
Title: Role of Esophageal Mast Cell Activation in Noncardiac Chest Pain (NCCP)
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21370
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Noncardiac Chest Pain (NCCP)
Keywords: NCCP, mast cell, esophagus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Chest pain is a common clinical complaint. About 30% patients with chest pain will have a normal coronary angiogram and are described as having noncardiac chest pain (NCCP). It is estimated that 25% of the population complain of chest pain at some time in their lifetime. The pathogenesis of NCCP is unknown. Esophageal hypersensitivity as a result of inflammation is considered to be an important mechanism in the development of this pain sensation. Little is currently known about the interaction between inflammatory mediators and peripheral afferent nerve terminals in the esophagus. The mast cell is one of the most enriched pro-inflammatory cells in the gastrointestinal tract. Activation of the mucosal mast cell releases a variety of mediators into adjacent tissues. We hypothesize that mediators released by mast cells sensitize esophageal nociceptors and induce pain sensation.

DETAILED DESCRIPTION:
1. Key Objectives: To determine the density and activation of esophageal mast cells in non-cardiac chest pain patients. We expect to find mast cell activation, as measured by mast cell count or degranluation, tryptase staining, and histamine release, will be greater in NCCP patients compared to controls, and the increased mast cell activation will correlate with the severity of NCCP. These results will expand our understanding of the pathogenesis of esophageal originated NCCP, and allow the development of new diagnostic and treatment options.
2. Study Population: (i) NCCP (ii) Reflux esophagitis (iii) Control subjects.
3. Summary of Procedures: (i) symptom assessment by chest pain questionnaire; (ii) esophageal reflux evaluation by review of records of 24-hour pH monitoring; (iii) evidence of esophagitis by endoscopy; (iv) esophageal biopsy by endoscopy; (v) mast cell activation study in biopsy specimen by mast cell count, tryptase and Transient receptor potential vanniloid-1 (TRPV1) staining, and histamine release assay.
4. Major Risks & Discomforts: There are no major risks & discomforts other than involved in standard upper GI endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* NCCP - presence of a history of chest pain with a negative cardiac evaluation, no evidence of gross esophagitis on endoscopy, and lack of any exclusion criteria; Reflux esophagitis - presence of chest pain or heartburn, negative cardiac evaluation, lack of exclusion criteria and presence of esophagitis on endoscopy;
* Controls - lack of history of chest pain, lack of exclusion criteria and lack of esophagitis on endoscopy. It is anticipated that patients being evaluated for heme positive stool or GI bleeding would be included as controls.

Exclusion Criteria:

- History of ischemic heart disease, history of asthma, significant food allergies, celiac disease, chronic inflammatory conditions (SLE, rheumatoid arthritis), atopic skin disease, varices, coagulopathy, recent drug treatment with steroids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-09; Primary Completion 2014-08-21 (Actual); Study Completion 2014-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaoyong Yu, MD, MPH, Principal Investigator — Department of Medicine, Penn State College of Medicine Hershey Medical Center; Ann Ouyang, MD, Study Director — Penn State College of Medicine Hershey Medical Center
Locations (1):
- Penn State College of Medicine Hershey Medical Center, Hershey, Pennsylvania, United States